CLINICAL TRIAL: NCT01131910
Title: Efficacy of TBE-vaccine to Patients With Rheumatic Disease Who Are Treated With Methotrexate and/or TNF-alfa Blocking Drugs
Brief Title: TBE-vaccine to Patients With Rheumatoid Arthritis Who Are Using Immunosuppressive Drugs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sormland County Council, Sweden (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Professor Lars Rombo, Sormland County Council
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2010-019438-28
Record Dates: First submitted 2010-05-24; First posted 2010-05-27 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2010-04

CONDITIONS: Rheumatoid Arthritis; Exposed to TBE-virus; Immunosuppression
Keywords: Rheumatoid arthritis; TBE-vaccine; Immunosuppression
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccination against TBE (Experimental): Less than 60 years old: Two doses of TBE- vaccine separated by a month and a third dose 12 months after the first dose
  60 years and above: Three doses, given at 0+1+3 months and a 4 th dose 12 months after the first dose
  Interventions: Biological: TBE-vaccine; Biological: Vaccination against TBE

INTERVENTIONS:
Biological: TBE-vaccine — Solution of 0.5 ml for intramuscular use. Given in 2 doses separated by 1 month to healthy individuals less than 60 years old. (3 doses 0+1+3 months to those are 60 and above in Sweden)
  Other Names: ATC-code J07B A01
Biological: TBE-vaccine — Solution for injection 0.5 ml im. 2 or 3 doses first years, 1 dose next year
  Other Names: J07B A01
Biological: Vaccination against TBE — 0.5 ml im at 0 and 1 month ( less than 60 years old) or 0 and 1 and 3 months (at least 60 years old)

SUMMARY:
The investigators intend to check whether the efficacy of a TBE-vaccine is substantially deteriorated in patients with rheumatoid arthritis who are treated with drugs which suppress the immune system. The investigators aim to detect a difference of at least 10 % compared to healthy individuals (historical controls) in protection when analysed with serology. If the investigators detect a difference, the investigators will continue to explore whether protection can be achieved by additional doses

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis treated with methotrexate and/or TNF-alfa blocking drugs
* Interest to be vaccinated
* Written consent
* Age 18 years or more

Exclusion Criteria:

* Previous TBE-infection
* Previous Vaccination with TBE
* Pregnancy
* Breast feeding
* Treatment with rituximab the last 9 months
* Inability to follow study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate | 1 year
  The humoral response to TBE-vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Lars Rombo, MD Professor, Principal Investigator — Somland county council
Locations (6):
- Dept infectious diseases, Helsingfors, Finland
- Sweden (5):
  - Dept infectious diseases, Eskilstuna
  - Dept. infectious diseases, Eskilstuna
  - Department of infectious diseases, Örebro
  - Department of infectious diseases, Stockholm
  - Dept infectious diseases, Uppsala